CLINICAL TRIAL: NCT05572632
Title: Community-based Pulmonary Rehabilitation (COPD Wellness) and Social Navigation (Health Advocates) to Improve Outcomes in Vulnerable Patients With COPD
Brief Title: Rehabilitation in Safety-net Environments (RISE) to Improve Outcomes in Vulnerable Patients With COPD
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21-35495; R01HL161049 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-10-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Social Needs; Chronic Disease; Health Disparities; Lung Diseases; Community Resources
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Wait-list randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The masked research coordinator will administer questionnaires and conduct clinical assessments at all study visits. Condition assignment will remain masked through data analysis and interpretation from study investigators and any team members involved in the data analysis. Furthermore, the COPD Wellness Coach leading weekly sessions, in addition to the research coordinator collecting endpoint measurements, will be masked to participant group status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPD Wellness (Experimental): This arm, COPD Wellness gives low-intensity exercise component with pulmonary rehabilitation for individuals with moderate-to-severe COPD. COPD Wellness is a program that was built from the Better Breathing Program, that is a part of San Francisco Health Network (SFHN) standard care for COPD.
  Interventions: Behavioral: COPD Wellness
- Usual Care (Active Comparator): This includes access to comprehensive primary care services. Participants randomized to the usual care arm will be offered referral to the Better Breathing Program that is part of SFHN standard care for COPD. This program consists of an evidence-based curriculum that improves disease knowledge and management skills but has no effect on symptoms or functional status. At end of study enrollment, usual care participants will be offered the COPD Wellness intervention.
  Interventions: Behavioral: Usual Care
- COPD Wellness Plus+ (Experimental): This arm includes COPD Wellness Plus+. This arm is built from COPD Wellness with the addition of Health Advocates (i.e. Plus+). This intervention seeks to understand the effects of addressing social needs on overall health and wellness through Zuckerberg San Francisco General Hospital's (ZSFG) Health Advocate (HA) program; participation and engagement with the HA's will serve as an adherence strategy.
  Interventions: Behavioral: COPD Wellness Plus+

INTERVENTIONS:
Behavioral: COPD Wellness — COPD Wellness consists of 10 weekly sessions led by the COPD Wellness Coach. The intervention was designed to be portable, rely on little equipment, and require limited space (~300sqft). The curriculum was iteratively developed with patient input and builds behavioral capability and self-efficacy through 30 minutes blocks of disease education and self-management skill building, exercise training, and social support.
  Arms: COPD Wellness
Behavioral: COPD Wellness Plus+ — Couples COPD Wellness with the ZSFG Health Advocates Program. The HA will help the participant prioritize identified needs and, using an algorithm informed approach to connect the individual to the needed resource, this includes providing referrals to outside social or legal service agencies, help with applications for social benefits, or other services. The HA will use a checklist to track activities including review and prioritization of needs, referrals or resources provided, and contacts/contact attempts.
  Arms: COPD Wellness Plus+
Behavioral: Usual Care — Includes access to comprehensive primary care services that is standardized across the SFHN. Participants randomized to the usual care arm will be offered referral to the Better Breathing Program that is part of SFHN standard care for COPD. At end of study enrollment, usual care participants will be offered the COPD Wellness intervention.
  Arms: Usual Care

SUMMARY:
Chronic obstructive pulmonary disease (COPD), one of the leading causes of death in the US, disproportionately affects low socioeconomic communities. While few interventions effectively modify the course of COPD and improve outcomes, pulmonary rehabilitation is the one notable exception. However, implementation of this resource-intensive program in real-life settings, and in particular, for underserved communities, has proven to be challenging. Safety-net centers that serve primarily under-insured populations lack financial resources to provide pulmonary rehabilitation.

The 10-week COPD Wellness and Plus+ Program directly addresses this gap, and yet, programs like these do not automatically lead to improved outcomes, which leads to the implementation of a Health Advocates program to address participant's social needs and barriers to healthcare.

DETAILED DESCRIPTION:
The proposed study will directly test the benefit of the 10-week COPD Wellness and Plus+ Program relative to usual care and estimate the added benefit of the HA in COPD Wellness Plus+ to COPD Wellness alone in a three-arm, randomized waitlist-controlled trial conducted in three geographically isolated urban primary care sites that provide care for some of the most socially vulnerable patient populations with COPD. In this Type 1 effectiveness-implementation hybrid design, the investigators aim to 1) determine the effectiveness of COPD Wellness and Plus+ to improve functional and symptom outcomes; and, using a mixed-methods approach 2) to evaluate the implementation of COPD Wellness and Plus+ across study sites applying the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) and Consolidated Framework for Implementation Research (CFIR) frameworks to identify additional barriers and enablers of intervention implementation and patient acceptance and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness to participate in the COPD Wellness program
* 40 to 90 years old
* English or Spanish speaking
* Physician-diagnosed COPD
* Spirometry-confirmed FEV1/FVC ratio <= 0.7 and FEV1% predicted <80% based on GLI-O prediction equation
* COPD Assessment Test ≥ 10 or history of 1+ exacerbation requiring hospitalization or 2+ outpatient exacerbations requiring steroid therapy
* Currently prescribed COPD medication(s)
* Ability to exercise with lower extremities
* No COPD exacerbations for ≥ 6 weeks
* Currently receiving care within SFHN

  * Note: Forced expiratory volume in the first second (FEV1); Forced vital capacity (FVC)

Exclusion Criteria:

* Pregnancy
* Dementia, cognitive impairment, or symptomatic psychiatric illness that would impair them from participating
* Unstable cardiovascular disease (includes recent [<6 months] myocardial infarction or pulmonary embolism, uncontrolled arrhythmia, poorly controlled heart failure)
* Other severe co-morbidity which means exercise is contraindicated (screened by Registered Nurse in consultation with Pulmonologist)
* Transmittable pulmonary infection (tuberculosis, COVID19)
* Participated in pulmonary rehabilitation in the past 12-months
* COPD exacerbation in the past 6 weeks
* Activities restrictions that limit one's ability to engage in moderate physical activity
* Other diagnosis or condition that carry a prognosis of death within the next year

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 6 Minute Walk Test to end-of-intervention (3-month) visit | 3-month (End of intervention) visit
  Standardized validated test to measure distance walked in 6 minutes

SECONDARY OUTCOMES:
Change from Baseline 6 Minute Walk Test at 6-month and 9-month visit following end-of-intervention | Baseline, 6-month, and 9-month visit following end-of-intervention
  Standardized validated test to examine functional status and measure distance walked in 6 minutes (reported in meters)
Change from Baseline COPD Assessment Test (CAT) at 3-month (End of Intervention) visit, 6-month, and 9-month visit | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Standardized validated comprehensive measure COPD Assessment Test (CAT) of symptom burden for individuals with COPD, minimum score: 0 - maximum score: 40, higher score indicates a more symptomatic COPD
Change from Baseline Quality of Life (SF-CRQ) assessment at 3-month (End of Intervention) visit, 6-month, and 9-month visit | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Health related quality of life is assessed using the validated Short-Form Chronic Respiratory Disease Questionnaire (SF-CRQ). This includes questions about four domains: dyspnea, fatigue, emotional function, and mastery. Items are answered using a 7-point scale Likert scale and summed within each domain. Higher results indicate a higher health-related quality of life.
Intervention Adherence at End-of-intervention (3 month) | Assessed during 10-week COPD Wellness Intervention
  Adherence as defined by the proportion of sessions attended out of ten
Change from Baseline COPD exacerbation history at 3-month (End of Intervention) visit, 6-month, and 9-month follow up | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Self-report non-standardized questionnaire on COPD exacerbation episodes; Exacerbation defined as a visit to an urgent care or emergency department for COPD, a hospitalization for COPD, or a prescription of an oral steroid for worsening COPD symptoms; not scored, higher exacerbations indicate more symptomatic COPD
Health System Proportion of patients referred to the intervention | Baseline, 24-months after study implementation
  Proportion of patients referred who enroll and participate in the study, which refers to the percent of patients referred that accept (attend 1+ session) COPD Wellness and Plus+ (intervention reach)
Health System Adoption of intervention for patients referred | Baseline, 24-months after study implementation
  Proportion of de novo referrals from primary care/post-hospitalization versus prompted referrals from research coordinator
Healthy System Maintenance of intervention from start of study to end of study activities | Baseline, Year 3 of study period (end of study activities)
  Referral pattern at start vs. at end of study period; staff and leadership intension to continue COPD Wellness and Plus+

OTHER OUTCOMES:
Change from Baseline Hospital Anxiety and Depression (HAD) Score at 3-month (End of Intervention) visit, 6-month, and 9-month visit | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  14-item standardized validated questionnaire titled Hospital Anxiety and Depression Scale (HADS) that includes sub-scales on anxiety and depression-- scores added at the end; minimum: 0 - maximum: 21; 0-7 is considered normal, 8-10 is considered borderline abnormal, 11-21 is considered abnormal
Change from Baseline Smoking Status at 3-month (End of Intervention) visit, 6-month, and 9-month visit | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Current use, duration of use, and pack-years will be assessed using the National Health Interview Survey (NHIS) Section IV Part A (Health Behaviors - Tobacco) questionnaire; standardized and validated; not scored
Change from Baseline Social Needs Screening at 3-month (End of Intervention) visit, 6-month, and 9-month follow up | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Using the Accountable Health Communities (AHC) Health Related Social Needs (HRSN) Screening Tool to assess for food and housing insecurity, transportation issues, and financial strain; standardized and validated; not scored, higher numbers indicate higher social need
Change in step count and accelerometry at 3-month (End of Intervention) visit, 6-month, and 9-month follow up | 3-month (End of intervention) visit, 6-month, and 9-month visit
  Step count and accelerometry as measured by FitBit Inspire 2 will be compared between the intervention groups (COPD Wellness & Plus+) and the waitlist control group, and between COPD Wellness and Plus+
Change in resting heart rate and heart rate variability at 3-month (End of Intervention) visit, 6-month, and 9-month follow up | 3-month (End of intervention) visit, 6-month, and 9-month visit
  Resting heart rate and heart rate variability as measured by Fitbit Inspire 2 will be compared between the intervention groups (COPD Wellness & Plus+) and the waitlist control group, and between COPD Wellness and Plus+
Change from Baseline Medication Adherence at 3-month (End of Intervention), 6-month, and 9-month visit | Baseline, 3-month (End of intervention) visit, 6-month, and 9-month visit
  Non-standardized validated questionnaire assessing mean number of days in which patient took all doses of controller medications (i.e., inhalers taken daily to prevent flare ups) as prescribed in last 7 days; seeking Electronic Health Record (EHR)-confirmation of healthcare visit (from COPD Exacerbation History) and medication prescription; not scored

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Thakur, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General (ZSFG) Hospital, San Francisco, California
  - Maxine Hall Health Center (MHHC), San Francisco, California
  - Southeast Health Center (SEHC), San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troosters T, Gosselink R, Decramer M. Short- and long-term effects of outpatient rehabilitation in patients with chronic obstructive pulmonary disease: a randomized trial. Am J Med. 2000 Aug 15;109(3):207-12. doi: 10.1016/s0002-9343(00)00472-1. PMID 10974183
- [Background] Baumann HJ, Kluge S, Rummel K, Klose H, Hennigs JK, Schmoller T, Meyer A. Low intensity, long-term outpatient rehabilitation in COPD: a randomised controlled trial. Respir Res. 2012 Sep 27;13(1):86. doi: 10.1186/1465-9921-13-86. PMID 23017153
- [Background] Selzler AM, Simmonds L, Rodgers WM, Wong EY, Stickland MK. Pulmonary rehabilitation in chronic obstructive pulmonary disease: predictors of program completion and success. COPD. 2012 Aug;9(5):538-45. doi: 10.3109/15412555.2012.705365. PMID 23030585
- [Background] Fischer MJ, Scharloo M, Abbink JJ, van 't Hul AJ, van Ranst D, Rudolphus A, Weinman J, Rabe KF, Kaptein AA. Drop-out and attendance in pulmonary rehabilitation: the role of clinical and psychosocial variables. Respir Med. 2009 Oct;103(10):1564-71. doi: 10.1016/j.rmed.2008.11.020. Epub 2009 May 29. PMID 19481919
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686